CLINICAL TRIAL: NCT00850070
Title: Sapropterin as a Treatment for Autistic Disorder: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Sapropterin as a Treatment for Autistic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Children's Health Council (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Glen R. Elliott, Chief Psychiatrist and Medical Director, The Children's Health Council
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHC-0901
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Autistic Disorder
Keywords: autism
MeSH Terms: conditions — Autistic Disorder | interventions — sapropterin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sapropterin, 100 mg capsules (Experimental): Sapropterin was supplied as a 100 mg tablet and dosage was based on 20 mg/kg/d, rounding to the nearest 100 mg. Most subjects crushed the tablets and administered it in liquid or a food to mask the taste. Subjects took the same dose daily for 16 weeks.
  Interventions: Drug: sapropterin
- Placebo, matching active drug (Placebo Comparator): The placebo was supplied as a 100 mg tablet, and dosage was based on 20 mg/kg/d, rounding to the nearest 100 mg. Most subjects crushed the tablets and administered it in liquid or a food to mask the taste. Subjects took the same dose daily for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sapropterin — Patients will receive sapropterin 20 mg per kilogram per day for 16 weeks
  Other Names: Kuvan; tetrahydrobiopterin
  Arms: sapropterin, 100 mg capsules
Drug: Placebo — Patients will receive a placebo identical in form and dosage to the active drug daily for 16 weeks.
  Other Names: sugar pill
  Arms: Placebo, matching active drug

SUMMARY:
This study is intended to provide a definitive test of the hypothesis that elevating sapropterin (tetrahydrobiopterin, a cofactor for several key brain enzymes)concentrations in the CNS will result in measurable improvements in core symptoms of autism in young individuals, under age 6 years. The study will entail a double-blind, placebo-controlled 16-week intervention.

DETAILED DESCRIPTION:
Over the past 20 years, several studies have suggested that sapropterin (tetrahydrobiopterin) might ameliorate core symptoms of autism at least in young (under age 6) subjects. However, those studies had somewhat questionable methodologies, a major one being that the doses of sapropterin used were roughly one tenth that thought to be needed to provide physiologically meaningful increases of sapropterin in the central nervous system (CNS). This study will look at the impact of a sustained exposure to this higher dose in well-diagnosed young children with autism.

ELIGIBILITY:
Inclusion Criteria:

* Parents sign informed consent
* Child meets criteria for autistic disorder (based on score on the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS), given by a certified administrator, research reliable)
* Child has a Developmental Quotient (DQ) ≥ 50 (Vineland Adaptive Scales, Interview Edition)
* Parents agree to delay initiation of other treatments during double-blind trial

Exclusion Criteria:

* Child has had seizures in past 6 months or a change in seizure medications in past 4 weeks.
* Child has > 18 points on subscale of (Autism Behavior Checklist) ABC-I
* Child is taking any psychoactive medication other than supplements, anticonvulsants, or soporifics (melatonin, diphenhydramine)
* Child has had any change in standing medications in the past 4 weeks.
* Child has known genetic disorders
* Child has known severe neurological disorders, including cerebral palsy

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glen R Elliott, Ph.D., M.D., Principal Investigator — The Children's Health Council
Locations (1):
- The Children's Health Council, Palo Alto, California, United States

REFERENCES:
- [Result] Klaiman C, Huffman L, Masaki L, Elliott GR. Tetrahydrobiopterin as a treatment for autism spectrum disorders: a double-blind, placebo-controlled trial. J Child Adolesc Psychopharmacol. 2013 Jun;23(5):320-8. doi: 10.1089/cap.2012.0127. PMID 23782126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment spanned from 4/09 to 6/11. A variety of methods were used to advertise the study, but most successful recruitment was word-of-mouth from study participants.
Pre-assignment Details: Few participants were excluded. Most common exclusions were failure to meet inclusion criteria, mostly absence of an autism diagnosis or cognitive functioning below the required minimum.
Groups:
- Sapropterin: tetrahydrobiopterin (BH4); dosage was 20mg/kg/day administered once per day orally in tablet form. Pills could be crushed and mixed with a variety of food substances (e.g., liquids or solids).
- Placebo: sugar pill; matched identical tablet, dosage was 20mg/kg/day administered once per day orally in tablet form. Pills could be crushed and mixed with a variety of food substances (e.g., liquids or solids).
Period: Overall Study
Arm/Group | Sapropterin | Placebo
Started | 23 | 23
Completed | 20 | 22
Not Completed | 3 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sapropterin: tetrahydrobiopterin (BH4)
- Placebo: sugar pill
- Total: Total of all reporting groups
Arm/Group | Sapropterin | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 23 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5 (1) | 5 (1) | 5 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 20 | 18 | 38
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression -- Improvement (CGI-I) Scale
Description: The CGI-I assessed the number of participants showing much or very much improvement on the CGI-I scale. This is a summary judgment made by a trained clinician based on observed and reported behaviors of the child compared to baseline. It is a 7-point scale from very much worse (1) to very much improved (7). Chi-square analyses were used to assess change in CHI-I scores (by group, post-test). Mixed-effects regression models via SPSS MIXED determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. We used random intercept and trend modeling that accounts for each individual's initial level of symptom severity/functioning and rate of change/time
Time Frame: Weekly for 4 weeks, then monthly, with 16-week end point. Primary outcome assessment used two time points, baseline and 16 weeks.
Population: This was an Intent-to-Treat Analysis with Last Observation Carried Forward.Analyses looked at percentage of children who improved (showing much or very much improved ratings) at 16-week time frame.
Measure: Number; unit: participants
Groups:
- Sapropterin: sapropterin 20 mg/kg/day
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
participants | 5 | 3
Statistical Analysis 1: Comparison: Sapropterin vs Placebo; Chi-square analyses were used to assess CGI-I scores. There were no transformations; Test type: Superiority or Other; p < .35, Chi-squared; Mean Difference (Final Values) = 2 — Estimated value comparison was active treatment minus placebo

2. Primary Outcome: Clinical Global Impression -- Severity (CGI-S) Scale
Description: The CGI-S assessed the number of participants with improved severity illness on the CGI-S scale. This is a summary judgment made by a trained clinician of symptom severity. It is a 7-point scale that rates the severity of the patient's illness at time of assessment with 1 - normal, not at all, to 7 - extremely ill. Mixed-effects regression models via SPSS MIXED determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. We used random intercept and trend modeling that accounts for each individual's initial level of symptom severity/functioning and rate of change/time
Time Frame: Baseline, 8 weeks, and 16 weeks. Primary outcome assessment used 2 time points, baseline and 16 weeks.
Population: This was an Intent-to-Treat Analysis with Last Observation Carried Forward.Analyses looked at number of children who improved (from markedly, severely or extremely ill to markedly, mildly or no illness) at 16-week time frame.
Measure: Number; unit: participants
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
participants | 3 | 1
Statistical Analysis 1: Comparison: Sapropterin vs Placebo; Test type: Superiority or Other; p < 0.06, Chi-squared; Mean Difference (Final Values) = 2

3. Secondary Outcome: Preschool Language Scale-Fourth Edition (PLS-4). Assesses Expressive and Receptive Language Skills in Ages Birth Through 6 Years, 11 Months.
Description: Measures expressive & receptive language and total scores in ages birth to 6 years 11 months. The scales generate raw, standard, and age-equivalent scores; raw scores for the total scale were selected for use in this study. Total is average of subscales. Minimum raw score = 0, maximum = 130. Higher scores indicate better language abilities. Mixed-effects regression models via SPSS MIXED determined the main effects attributed to differences by group (BH4 and placebo), time (treated as categorical at levels baseline, 8 weeks, and 16 weeks) and the group-by-time interaction. For the outcome effect, the difference between baseline and 16 weeks was determined as an indicator for change.
Time Frame: Primary outcome assessment examined the difference in scores between baseline and week 16.
Population: Intent-to-treat analysis; all subjects included. Difference in scores between baseline and 16 weeks was used as treatment outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 84 (29) | 60 (25)

4. Secondary Outcome: Vineland Adaptive Behavior Scale-II.
Description: the Vineland-2 is a semi-structured interview designed to assess communicatino, daily living, socialization and motor skills. The Vineland-2 is comprised of a total Adaptive Composite scale; we chose to use 10 subscales that specifically address functional domains relevant for a young ASD sample - Receptive Communication, Expressive Communication, Personal Daily Living Skills, Domestic Daily Living Skills, Community Daily Living Skills, Interpersonal Relations, Play Skills, Coping Skills, Gross Motor Skills, Fine Motor Skills. Scales generate raw or sum, V-, and age-equivalent scores; raw scores were selected for use in the study. Raw score ranges from 0 to 108 depending on the scale. Total raw scale range is from 0 to 766. Subscale scores are averaged to create the total adaptive behavior composite. Higher subscale scores indicate more skills. Difference between baseline and week 16 was used as an indicator of change.
Time Frame: Primary outcome assessment used two time points, baseline and 16 weeks.
Population: Intent-to-treat analysis; all subjects included. Includes mean at 16-week outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 344.76 (50.0) | 294.9 (70.1)

5. Secondary Outcome: Children's Yale Brown Obsessive Compulsive Scale (C-YBOCS)
Description: The C-YBOCS is a scale is designed to rate the severity of obsessive and compulsive symptoms in children and adolescents, ages 6 to 17 years. It can be administered by a clinican or trained interviewer in a semi-structured fashion. In general, the ratings depend on the child's and parent's report; however, the final rating is based on the clinical judgement of the interviewer. Rate the characteristics of each item over the prior week up until, and including, the time of the interview. Scores should reflect the average of each item for the entire week, unless otherwise specified.
Time Frame: Baseline, 8 weeks, and 16 weeks
Population: The data was not analyzed secondary to lack of significant findings in the primary outcome measure. Also, limited data collected secondary to the age range of the children we saw.The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Sapropterin, 100 mg Capsules | Placebo, Matching Active Drug
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Connor's Preschool ADHD Questionnaire
Description: Conners Early Childhood, addresses child behavior for ages 2 years to 6 years with a variety of scales, including an ADHD subdomain.
Time Frame: Baseline, 8 weeks, and 16 weeks
Population: Data was not analyzed secondary to lack of significant findings in primary outcome measures and limited data collected on this instrument. The data cannot now be provided as the research team has since disbanded and it is not possible to reanalyze the data at this time.
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Adverse Events Scale
Description: This was not a standardized scale but a set of questions that was asked of each family - some standard and others open ended.
Time Frame: Every 1-2 weeks for 16 weeks
Population: We did not specifically analyze this data but instead use it as a guide to determine if a drug should be discontinued for a particular child.
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Aberrant Behavior Checklist (ABC) - Inappropriate Speech
Description: Subscale assessing echolalia & other odd speech. Higher subscale scores indicate more symptoms. 4 items comprise the subscale, with range of scores from 0-4. Total score range on this subscale is 0 to 16. Scores are averaged to compute overall score. Difference in scores between baseline and week 16 were used as indicator of change.
Time Frame: Primary outcome assessment used two time points, baseline and 16 weeks.
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 2.6 (1.9) | 3.9 (3.6)
Statistical Analysis 1: Comparison: Sapropterin vs Placebo; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -2, Standard Error of Mean 0.9

9. Secondary Outcome: Social Responsiveness Scale (SRS)
Description: The SRS is a 65-item scale used to measure the severity of symptoms in ASD as they occur in natural social settings. The SRS is comprised of 1 Total scale and 5 subscales that generate raw scores that can be converted to standard T-scores (with mean of 50 and standard deviation of 10) for gender and rater type; standard scores were selected for use in this study. A total T-score of 76 or higher is considered severe and strongly associated with a clinical diagnosis of autistic disorder. A t-score of 60-75 is in the mild to moderate range and considered typical for children with mild or 'high-functioning' ASD, while a T-score of 59 or less suggests an absence of ASD symptoms. A total raw score of >75 were associated with a sensitivity value of .85 and a specificity value of .75 for ASD. Difference in scores between baseline and week 16 were used as an indicator of change.
Time Frame: Primary outcome assessment used two time points, baseline and 16 weeks.
Population: Intent-to-treat analysis; all subjects included. Includes mean at 16-week outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale | 76.7 (10.9) | 83.2 (10.4)

10. Secondary Outcome: Parent Global Assessment (PGA) Scale
Description: This is a measure where parents rate their impression of their child's improvement, in a global manner.
Time Frame: Baseline, 8 weeks, and 16 weeks
Population: as for outcome 6
Arm/Group | Sapropterin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for the length of the study, i.e., 16 weeks.
Arm/Group | Sapropterin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/23
Other Adverse Events (participants affected / at risk) | 10/23 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin (N=23) | Placebo (N=23)
transient viral rash (Skin and subcutaneous tissue disorders) | 2 | 0 — Viral or autoimmune rashes
seizure disorder (Nervous system disorders) | 0 | 1 — New-onset seizures
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin (N=23) | Placebo (N=23)
irritablity (Psychiatric disorders) | 5 | 4 — Increased irritablility in a variety of settings
difficulty sleeping (Nervous system disorders) | 2 | 4 — Persistent changes in sleep, including onset insomnia, frequent wakening during the night, lightening of sleep
Change in Bowel Habits (Gastrointestinal disorders) | 0 | 4 — Changes in stool consistency or bowel movement frequency
repetitive behaviors (Nervous system disorders) | 1 | 2 — Sustained changes in or appearance of stereotypies or other odd, repetitive behaviors
hyperactivity (Nervous system disorders) | 2 | 1 — Persistent increase in overall activity level in a variety of settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No